CLINICAL TRIAL: NCT02538289
Title: Hospital Without Dyspnea. Rationale and Design of a Multidisciplinary Intervention
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital General Universitario Gregorio Marañon (Other)
Collaborators: Instituto de Salud Carlos III (Other Government)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Hospital without dyspnea
Record Dates: First submitted 2015-08-31; First posted 2015-09-02 (Estimated); Last update posted 2017-02-24 (Actual); Status verified 2016-02

CONDITIONS: Dyspnea
Keywords: Dyspnea; Palliative Care; Heart Failure; Chronic Pulmonary Disease; Opioids
MeSH Terms: conditions — Dyspnea; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Patients admitted before talks (Other): Patients admitted to Cardiology or Respiratory Medicine Departments before the interventional teaching talks.
  Interventions: Behavioral: Teaching talks
- Patients admitted after talks (Other): Patients admitted to Cardiology or Respiratory Medicine Departments after the interventional teaching talks.
  Interventions: Behavioral: Teaching talks

INTERVENTIONS:
Behavioral: Teaching talks — Two teaching talks specifically addressed to medical staff which concerns the adequate treatment and needs of dyspneic patients, including pharmacological and non-pharmacological treatment.

SUMMARY:
Dyspnea is a symptom that is growing in incidence, as respiratory and heart diseases are becoming more frequent. Patients suffering from dyspnea have a significant disabling due to chronic refractory dyspnea and crisis of irruptive dyspnea. Although there are several tools that may produce an improvement of symptom intensity, they are underused.

DETAILED DESCRIPTION:
We sought to investigate whether if teaching interventions specifically addressed to medical staff improve the well-being of dyspneic patients. The MAIN GOAL of this study is to evaluate the effect of two talks (conveyed to doctors and nurses of Cardiology and Respiratory Medicine Departments) on the patient-perceived dyspnea. The contents of these talks will be prepared and supervised by Palliative Care specialists.

This is a four-staged study that includes a first observational phase (prevalence study of dyspnea) followed by intervention and a third phase that will determine the effect of this teaching intervention. The fourth phase consists in the elaboration of specific protocols for management of dyspnea.

A pharmacovigilance study of opioids will also take place.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission with dyspnea as main symptom
* Acceptance of participation in the study
* Diagnosis of Chronic Respiratory Disease
* Diagnosis of Chronic Heart Failure
* Chronic Refractory Dyspnea higher than 1/10 and Irruptive Dyspnea higher than 2/10 degree by Rating Numerical Scale

Exclusion Criteria:

* Cognitive Impairment
* Voluntary dropout.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2016-04 (Actual); Primary Completion 2017-09 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Decrease the number of patients with advanced heart or chronic respiratory diseases who present chronic refractory dyspnea or irruptive dyspnea and do not receive adequate treatment. | One month
  Decrease the number of patients admitted to Cardiology or Respiratory Medicine departments who present chronic respiratory dyspnea or irruptive dyspnea.

SECONDARY OUTCOMES:
Detect the prevalence of dyspnea in patients admitted to our hospital. | One month
  Number of patients.
Describe the therapeutic tools (pharmacological and no pharmacological) employed for symptomatic treatment of dyspnea. | One month
  Frequency of methods usage for dyspnea relief.
Evaluate the impact on dyspnea intensity associated with an implementation of educational talks addressed to medical staff in the management of dyspnea. | One year
  Numerical Rating Scale score.
Number of patients that continue chronic treatment with opioids for chronic refractory dyspnea and irruptive dyspnea. | Three months
  Number of patients that receive opioid treatment at three months of inclusion
Determine the intensity and functional impact of dyspnea in patients admitted to our hospital. | One month
  Dyspnea intensity by Numerical Rating Scale score
Determine the efficacy derived from a chronic treatment with opioids for chronic refractory dyspnea and irruptive dyspnea. | Three months
  Dyspnea intensity by Numerical Rating Scale score
Determine the number of patients that present side effects derived from a chronic opioid treatment that require lowering dose or stopping treatment. | Three months
  Number of patients that present side effects
Determine whether a specific educational talk would be affordable for dyspnea management | One month
  Costs in euros invested in medical staff training

CONTACTS AND LOCATIONS:
Overall Officials: Juan Manuel Nuñez Olarte, M.D., Principal Investigator — Hospital General Universitario Gregorio Marañon
Locations (1):
- Gregorio Marañon University Hospital, Madrid, Madrid, Spain

REFERENCES:
- [Background] Badia X, Muriel C, Gracia A, Nunez-Olarte JM, Perulero N, Galvez R, Carulla J, Cleeland CS; Grupo Vesbpi. [Validation of the Spanish version of the Brief Pain Inventory in patients with oncological pain]. Med Clin (Barc). 2003 Jan 25;120(2):52-9. doi: 10.1016/s0025-7753(03)73601-x. Spanish. PMID 12570914